CLINICAL TRIAL: NCT06901960
Title: Monitoring Hyperkalemia Using Point-of-care AI-enabled ECG Device Among Patients With Chronic Kidney Disease Stages 3b-5 to Reduce Rate of Hyperkalemia - a Practical Randomized Clinical Trial
Brief Title: Monitoring Hyperkalemia Using Point-of-care AI-enabled ECG Device Among Patients With Chronic Kidney Disease Stages 3b-5
Acronym: POCKET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-943
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease (Stages 3b-5)
Keywords: Chronic kidney disease; hyperkalemia; ECG
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperkalemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitoring plasma potassium using ECG device (Experimental): Patients in this arm will use AI-enhanced point-of-care ECG device to monitor their serum potassium level every 3 days for 6 months in addition to their regular outpatients follow-up. If ECG device detected hyperkalemia was reported, more intensive monitoring, education on diet or offer of making outpatient appointment, as appropriate, will be provided.
  Interventions: Device: A mobile artificial intelligence-enhanced electrocardiogram device estimating plasma potassium categories (<5 mmol/L, 5 - <5.5 mmol/L, 5.5 - <6.0 mmol/L and ≥ 6.0 mmol/L)
- Regular outpatients follow-up (No Intervention): Patients in this arm will just follow their regular outpatients care without additional intervention.

INTERVENTIONS:
Device: A mobile artificial intelligence-enhanced electrocardiogram device estimating plasma potassium categories (<5 mmol/L, 5 - <5.5 mmol/L, 5.5 - <6.0 mmol/L and ≥ 6.0 mmol/L) — A mobile AI-enhanced electrocardiogram device will be used to help patients monitor hyperkalemia. The device, shaped like a stick of chewing gum, collects time-series data of electrocardiogram lead I through two electrodes. Deep convolutional neural network algorithm can read the data and generated categories of plasma potassium (<5 mmol/L, 5 - <5.5 mmol/L, 5.5 - <6.0 mmol/L and ≥ 6.0 mmol/L). Study participants receive the device after randomization. The staff establishes a WeChat group for each participant and reminds them to monitor plasma potassium every 3 days. When the detected plasma potassium category falls in 5 - <5.5 mmol/L, they will be reminded to watch diet and to verify plasma potassium again. More intensive reminding (once daily) will be sent if plasma potassium category falls in 5.5 - <6.0 mmol/L or ≥ 6.0 mmol/L. An extra outpatient appointment will also be made as soon as possible for the patients when their detected plasma potassium category is ≥ 6.0 mmol/L.
  Arms: Monitoring plasma potassium using ECG device

SUMMARY:
The clinical trial will be conducted in a real-world outpatients setting with the goal of learning if monitoring serum potassium frequently among patients with moderate-to-advanced stages of chronic kidney disease leading to optimal management of hyperkalemia (the reduced occurrence of serum potassium ≥ 5.0 mmol/L during 6 months of follow-up). It will also learn about the adherence of using a mobile monitoring device.

Participants will:

* Measure their serum potassium using an AI-enhanced point-of-care ECG device at least twice per week
* Receive health education prompts to reduce intake of potassium rich foods if their electrocardiogram device measured serum potassium is abnormal
* Receive alerts to visit nephrology clinic if their electrocardiogram device measured serum potassium is continuously abnormal

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease stages 3b-5 (eGFR: 10 - <45 ml/min/1.73m²)
* Patients with regular visits in the study sites to manage their chronic kidney disease (≥ 1 visit per 3 months during the past year before enrollment)
* Willingness to participate in the study with signed informed consent

Exclusion Criteria:

* Patients already under kidney replacement therapy or will receive kidney replacement therapy in 6 months
* Unwillingness or without the ability to monitor hyperkalemia using the study device
* Patients with heart pacemaker implanted

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1066 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of serum potassium ≥ 5.0 mmol/L | Six months (+1 month if outpatients visit delayed) after enrollment into the study
  The serum potassium should be the laboratory measured one, which is obtained in the 3(±1) month and 6(±1) month follow-up in outpatients visit.

SECONDARY OUTCOMES:
Average level of serum potassium | Six month (+1 month if outpatients visit delayed) after enrollment into the study
  The serum potassium should be the laboratory measured one, which is obtained in the 3(±1) month and 6(±1) month follow-up in outpatients visit.
Frequency of using AI-enhanced ECG device to monitor serum potassium | Six months (+1 month if outpatients visit delayed) after enrollment into the study and 3 months (+1 month if outpatients visit delayed) after the 6 months of intervention.
  The frequency will be monitored in intervention period for the intervention group and after intervention (up to 4 months) for both the original intervention and control groups.

OTHER OUTCOMES:
Incidence of serum potassium ≥ 5.0 mmol/L after the intervention period | Three months (+1 month if outpatients visit delayed) after the 6 months of intervention
  We collect incidence of serum potassium ≥ 5.0 mmol/L after the intervention period to see whether there is still a gap between the original intervention and control groups with the latter one having obtained the device.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Hubei Provincial Hospital of TCM, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication will be shared upon reasonable request.